CLINICAL TRIAL: NCT07399561
Title: A Randomized Controlled Trial Evaluating the Effects of Exercise on Chemotherapy-Induced Peripheral Neuropathy in Patients Treated With Oxaliplatin or Paclitaxel
Brief Title: Effect of Exercise on Chemotherapy-Induced Peripheral Neuropathy
Acronym: EX-CIPN
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: National Cancer Center, Korea (Other Government)
Responsible Party: Principal Investigator, Su-hyun Kim, Head of Department of Neurology, National Cancer Center, Korea
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: NCC-CIPN-EX-2025
Record Dates: First submitted 2026-01-18; First posted 2026-02-10 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Peripheral Neuropathy, Secondary to Drugs or Chemicals; Oxaliplatin Induced Peripheral Neuropathy in Cancer Patients; Paclitaxel Induced Neuropathy
Keywords: chemotherapy induced peripheral neuropathy; CIPN; Exercise
MeSH Terms: conditions — Peripheral Nervous System Diseases; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Exercise Intervention (Experimental): Participants assigned to this arm will perform a structured home-based exercise program during chemotherapy and for up to three months after completion of chemotherapy. The exercise program is designed to be safe and feasible during active cancer treatment and includes aerobic and strengthening components. Participants receive standardized exercise education materials, and adherence and safety are monitored through regular telephone follow-up.
  Interventions: Behavioral: Exercise Intervention
- Usual Care (Active Comparator): Participants assigned to this arm will receive standard oncologic care and general education regarding chemotherapy-induced peripheral neuropathy. No structured exercise program is prescribed during the study period.
  Interventions: Other: Usual Care

INTERVENTIONS:
Behavioral: Exercise Intervention — A structured home-based exercise program performed during chemotherapy and for up to three months after completion of chemotherapy. The program includes aerobic and strengthening exercises and is designed to be safe and feasible during active cancer treatment. Adherence is monitored through regular telephone follow-up.
  Arms: Exercise Intervention
Other: Usual Care — Standard oncologic care and general education regarding chemotherapy-induced peripheral neuropathy, without a structured exercise program.
  Arms: Usual Care

SUMMARY:
Chemotherapy-induced peripheral neuropathy (CIPN) is a common and often persistent adverse effect of oxaliplatin- and paclitaxel-based chemotherapy. While exercise is frequently recommended for patients with CIPN, it remains unclear whether exercise mitigates neuropathic injury itself or primarily improves physical function and quality of life.

This randomized controlled trial evaluates the effects of exercise on CIPN during and after chemotherapy. Patients receiving oxaliplatin for colorectal cancer or paclitaxel for gynecologic cancer are randomized to an exercise intervention or usual-care control. Neuropathy severity is assessed using objective neurophysiological measures, blood biomarkers, and validated clinical and patient-reported outcomes.

DETAILED DESCRIPTION:
This is an open-label, randomized controlled trial conducted in patients undergoing neurotoxic chemotherapy. Two chemotherapy cohorts are included: patients receiving oxaliplatin-based chemotherapy for colorectal cancer and patients receiving paclitaxel-based chemotherapy for gynecologic cancer.

Participants are randomized 1:1 to an exercise intervention group or a usual-care control group. Randomization is performed prior to chemotherapy initiation, with stratification by age group and chemotherapy regimen to ensure balance between groups.

The exercise intervention consists of a structured home-based exercise program initiated at the start of chemotherapy and continued until three months after completion of chemotherapy. The program is designed to be safe and feasible during active cancer treatment, with adherence monitored through regular follow-up.

The primary objective is to determine whether exercise reduces the severity of chemotherapy-induced peripheral neuropathy, as assessed by objective neurophysiological testing and validated patient-reported measures. Secondary objectives include evaluation of blood biomarkers of neuroaxonal injury and inflammation, physical function, and quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of colorectal cancer (oxaliplatin cohort) or gynecologic cancer (paclitaxel cohort)
* Planned initiation of oxaliplatin- or paclitaxel-based chemotherapy
* Karnofsky Performance Status ≥70
* Ability to provide written informed consent

Exclusion Criteria:

* Pre-existing peripheral neuropathy from other causes
* Severe comorbidities limiting safe participation in exercise
* Regular participation in a structured moderate- to high-intensity exercise program comparable to the study intervention prior to enrollment.
* Cognitive impairment interfering with study participation

Ages: 19 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Estimated)
Dates: Start 2026-02-03 (Estimated); Primary Completion 2027-07-01 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in Chemotherapy-Induced Peripheral Neuropathy Severity (CTCAE v5.0) | Baseline (prior to initiation of chemotherapy), end of chemotherapy (up to approximately 24 weeks after chemotherapy initiation), and 3 months after completion of chemotherapy.
  Change in chemotherapy-induced peripheral neuropathy severity assessed using the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI-CTCAE) version 5.0 sensory neuropathy grade (Grade 0-4, with higher grades indicating more severe neuropathy).

SECONDARY OUTCOMES:
Blood Biomarkers | Baseline, end of chemotherapy, 3 months post-chemotherapy
  Serum neurofilament light chain (NfL), brain-derived neurotrophic factor (BDNF), nerve growth factor (NGF), complement components (e.g., C5a), and inflammatory cytokines.
Quality of Life Assessed by EORTC QLQ-C30 | Baseline, end of chemotherapy (up to approximately 24 weeks), and 3 months after completion of chemotherapy.
  Quality of life assessed using the European Organisation for Research and Treatment of Cancer Quality of Life Questionnaire-Core 30 (EORTC QLQ-C30). The questionnaire generates scores ranging from 0 to 100. For the global health status and functional scales, higher scores indicate better quality of life and functioning, whereas for symptom scales, higher scores indicate greater symptom burden.
Change in Timed Up and Go Test Performance | Baseline (prior to initiation of chemotherapy), end of chemotherapy (up to approximately 24 weeks after chemotherapy initiation), and 3 months after completion of chemotherapy.
  Change in mobility and balance assessed using the Timed Up and Go (TUG) test, measured in seconds, with longer times indicating poorer performance.
Change in Sensory Nerve Action Potential Amplitude | Baseline (prior to initiation of chemotherapy), end of chemotherapy (up to approximately 24 weeks after chemotherapy initiation), and 3 months after completion of chemotherapy.
  Change in sensory nerve action potential (SNAP) amplitude of predefined sensory nerves assessed by nerve conduction studies, measured in microvolts (µV), with lower amplitudes indicating greater axonal dysfunction.
Change in Patient-Reported CIPN Symptoms Assessed by EORTC QLQ-CIPN20 | Baseline, end of chemotherapy (up to approximately 24 weeks), and 3 months after completion of chemotherapy.
  Change in chemotherapy-induced peripheral neuropathy symptoms assessed using the European Organisation for Research and Treatment of Cancer Quality of Life Questionnaire-Chemotherapy-Induced Peripheral Neuropathy 20-item scale (EORTC QLQ-CIPN20; score range 0-100, with higher scores indicating worse neuropathy).
Change in Serum Neurofilament Light Chain Concentration | Baseline (prior to initiation of chemotherapy), end of chemotherapy (up to approximately 24 weeks after chemotherapy initiation), and 3 months after completion of chemotherapy.
  Change in serum neurofilament light chain (NfL) concentration, a biomarker of neuroaxonal injury, measured using a validated immunoassay.
Change in Serum Brain-Derived Neurotrophic Factor Level | Baseline, end of chemotherapy (up to approximately 24 weeks), and 3 months after completion of chemotherapy.
  Change in serum brain-derived neurotrophic factor (BDNF) level, measured using a single molecule array (SIMOA) immunoassay.
Change in Serum Complement Component C5a Level | Baseline (prior to initiation of chemotherapy), end of chemotherapy (up to approximately 24 weeks after chemotherapy initiation), and 3 months after completion of chemotherapy.
  Change in serum complement component C5a level, a marker of complement activation, measured using the MicroVue™ C5a enzyme immunoassay.
Change in Sit-to-Stand Test Performance | Baseline, end of chemotherapy (up to approximately 24 weeks), and 3 months after completion of chemotherapy.
  Change in lower extremity functional strength assessed using the Sit-to-Stand test, measured as time to complete the test or number of repetitions, as applicable.
Change in 2-Minute Walk Test Distance | Baseline, end of chemotherapy (up to approximately 24 weeks), and 3 months after completion of chemotherapy.
  Change in functional exercise capacity assessed using the 2-Minute Walk Test, measured as total distance walked in meters.
Change in Handgrip Strength | Baseline, end of chemotherapy (up to approximately 24 weeks), and 3 months after completion of chemotherapy.
  Change in upper extremity muscle strength assessed using handgrip dynamometry, measured in kilograms, with lower values indicating reduced strength.
Secondary Outcome: Sensory Nerve Conduction Velocity | Baseline (prior to initiation of chemotherapy), end of chemotherapy (up to approximately 24 weeks after chemotherapy initiation), and 3 months after completion of chemotherapy.
  Change in sensory nerve conduction velocity of predefined sensory nerves assessed by nerve conduction studies, measured in meters per second (m/s), with lower velocities indicating greater demyelination or conduction slowing.
Change in Serum Nerve Growth Factor Level | Baseline, end of chemotherapy (up to approximately 24 weeks after chemotherapy initiation), and 3 months after completion of chemotherapy.
  Change in serum nerve growth factor (NGF) level, measured using a validated immunoassay.
Change in Circulating Inflammatory Cytokine Levels | Baseline, end of chemotherapy (up to approximately 24 weeks), and 3 months after completion of chemotherapy.
  Change in circulating levels of selected pro- and anti-inflammatory cytokines measured using a multiplex enzyme-linked immunosorbent assay.

CONTACTS AND LOCATIONS:
Locations (1):
- National Cancer Center, Goyang, Gyeonngi, South Korea

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data underlying the results reported in the manuscript.
Supporting Information: Study Protocol, SAP
Time Frame: Beginning 6 months after publication of the primary results and ending 5 years after publication.
Access Criteria: Individual participant data will be shared upon reasonable request. Requests must include a methodologically sound proposal and be approved by the study investigators. Data will be shared after execution of a data sharing agreement, in accordance with institutional policies and applicable regulations.